CLINICAL TRIAL: NCT03272334
Title: A Phase I/II Study of Anti-CD3 X Anti-HER2/neu (Her2Bi) Armed Activated T Cells (ATC) and Pembrolizumab Combination Therapy in Women with Metastatic Breast Cancer
Brief Title: Her2-BATS and Pembrolizumab in Metastatic Breast Cancer
Acronym: Breast-47
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Patrick Dillon, MD, Assistant Professor, Hematology and Oncology, University of Virginia
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19406
Record Dates: First submitted 2017-08-28; First posted 2017-09-05 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; Adoptive Cell Therapy; Armed Activated T-cells; Bispecific Antibodies; Immunotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Pembrolizumab administered in combination with HER2 Bispecific Antibody Armed Activated T-Cell (BATs) infusions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Schedule #1 (Experimental): At approximately 4 weeks following leukapheresis, 8 infusions of HER2 BATs are given twice weekly in weeks #1, #2, #5, and #6 plus 1 infusion of Pembrolizumab in week #7. No interventions within weeks #3 and 4.
  Interventions: Drug: HER2 BATs with Pembrolizumab
- Schedule #2 (Experimental): At approximately 4 weeks following leukapheresis, 8 infusions of HER2 BATs are given twice weekly in weeks #1, #2, #5, and #6 plus 2 infusions of Pembrolizumab; the first given within weeks #3 - 4 and the second in week #7.
  Interventions: Drug: HER2 BATs with Pembrolizumab
- Schedule #3 (Experimental): At approximately 4 weeks following leukapheresis, 8 infusions of HER2 BATs are given twice weekly in weeks #1, #2, #5, and #6 plus 3 infusions of pembrolizumab; the first given one week prior to first BATs infusion, the second is given within weeks #3 - 4, and the third at week #7.
  Interventions: Drug: HER2 BATs with Pembrolizumab

INTERVENTIONS:
Drug: HER2 BATs with Pembrolizumab — 8 infusions of HER2 BATs with 1-3 infusions of Pembrolizumab

SUMMARY:
This proposal uses HER2Bi armed activated T-cells (HER2 BATs) to target breast cancer in combination with pembrolizumab (PBZ) in women with metastatic breast cancer (MBC). Phase I will determine a safe dose of the combination of PBZ and HER2 BATs in 3 to 18 patients. In the phase II portion, an additional 12 patients will be treated at the selected dose to further evaluate the safety and preliminary efficacy.

Study treatment includes a combination of 8 infusions of BATs using a previously established schedule and one to three infusions of PBZ (200 mg per dose). PBZ will be added to 8 infusions of BATs in 3 schedules: #1) after the 8th BATs infusion; #2) after the 4th and 8th BATs infusions; and then, #3) before the 1st and after the 4th and 8th BATs infusions.

DETAILED DESCRIPTION:
Once subjects are determined eligible, white blood cells (lymphocytes) are collected via leukapheresis procedure. Depending on arm/schedule, about 4-5 weeks later, study treatment will begin. For HER2 BATs, the white blood cells, specifically T cells, are then mixed with two proteins - OKT3 and IL-2 -- which activates the cells to multiply. After approximately 14 days in culture, the activated T cells are coated with OKT3 and trastuzumab/Herceptin (HER2Bi), and washed to remove excess Herceptin in order to produce bispecific antibody armed T cells (BATs). Cells are then frozen and stored until scheduled to be infused.

Follow-up appointment schedule will include clinic visits 2 weeks, 1 month, 3 months, and 6 months after the last dose of Pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed breast cancer (infiltrating ductal or lobular breast carcinoma) with evidence of measurable metastatic disease. Metastatic disease must be biopsy proven.

   a. Since histologic type, lymphatic permeation, blood vessel invasion, and degree of anaplasia may be prognostic variables, appropriate slides of the primary lesion will be requested for future review. HER2, estrogen, and progesterone receptor positivity will be recorded.
2. Measurable lesion. Patients are required to have at least one measurable non-bone lesion ≥10 mm that has not been irradiated.

   a. Measurable metastatic disease documented by radiograph, CT scan, PET/CT, MRI, or physical exam is required. Each subject will be required to have at least one measurable lesion that has not been irradiated with a minimum size in at least one diameter of ≥ 10 mm for liver lesions, lung, skin, and ≥ 15 mm lymph node metastases. Biopsy of recurrent site(s) is not required.
3. Patients must have HER2 status determined by FISH or IHC. HER2 status of positive or negative are both eligible for the study.

   In order to be eligible for participation in this trial, the patient must also:
4. Be female ≥ 18 years of age
5. Be willing and able to provide written informed consent for the trial.
6. Have a performance status (PS) ECOG 0-1
7. Have a life expectancy ≥ 3 months
8. Be eligible for apheresis, as determined by the Stem Cell Transplant team
9. Demonstrate adequate organ function as defined below, all screening labs should be performed within 10 days prior to apheresis.

   Absolute lymphocyte count ≥ 500/mm3 Absolute neutrophil count (ANC) ≥1,500 /mcL Platelets ≥ 100,000 / mcL Hemoglobin ≥ 9 g/dL (or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment) BUN ≤ 1.5 X upper limit of normal (ULN) Serum creatinine OR ≤1.5 X upper limit of normal (ULN) OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN Serum total bilirubin ≤ 1.5 X ULN OR AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases Albumin >2.5 mg/dL International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy Activated Partial Thromboplastin Time (aPTT) as long as PT or PTT is within therapeutic range of intended use of anticoagulants
10. Female patients of childbearing potential should have a negative urine or serum pregnancy test at screening. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
11. Female patients of childbearing potential must be willing to use an adequate method of contraception as outlined in Section 4.5.2, for the course of the study through 120 days after the last dose of study medication.
12. Patients must have had two or more lines of prior therapy (chemo or hormonal) in the metastatic setting

Exclusion Criteria:

The patient must be excluded from participating in the trial if the subject:

1. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to leukapheresis.
2. Has a known history of active TB (Bacillus Tuberculosis)
3. Hypersensitivity to PBZ or any of its excipients.
4. Lack of recovery (i.e., ≤ Grade 1 or baseline prior to last line of cancer therapy) from non-laboratory adverse events except ≤ Grade 2 neuropathy
5. Has history of another malignancy within the past 5 years. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
6. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to leukapheresis. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
7. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
8. Has known history of, or any evidence of active, non-infectious pneumonitis.
9. Has an active infection requiring systemic therapy.
10. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
11. Is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
12. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
13. Has Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies) or known history of Hepatitis B (e.g., HBsAg reactive) or Hepatitis C antibody is detected. Note: Patients may be eligible if HCV antibody is detected as long as HCV viral load is undetectable following an FDA approved treatment regimen
14. Has received a live vaccine within 30 days of apheresis. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
15. Has a history of significant cardiac disease, including:

    * History of a recent myocardial infarction (within one year), a past myocardial infarction (more than one year ago) along with current coronary symptoms requiring medications and/or evidence of depressed left ventricular function (LVEF < 45% by MUGA or ECHO).
    * Current history of angina/coronary symptoms requiring medications and/or evidence of depressed left ventricular function (LVEF < 45% by MUGA or ECHO)
    * Clinical evidence of congestive heart failure requiring medical management (irrespective of ECHO results).
16. Pt may be excluded if, in the opinion of the PI and investigator team, the pt is not capable of being compliant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2017-12-29 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities on each schedule/arm | The study will not advance to the next schedule until 3 weeks after the last patient in the cohort completes her last dose of Pembrolizumab.
  Maximum tolerated dose will be based on number of dose limiting toxicities in each schedule/arm

SECONDARY OUTCOMES:
Dose Limiting Toxicities on the selected arm in the expansion cohort | All dose limiting toxicities are expected to be identified within the three weeks following the last dose of Pembrolizumab
  Dose Limiting toxicities on the arm selected based on the dose/schedule selection part of the study. More patients will be enrolled onto this cohort to confirm safety.
Immune response to treatment in blood | Blood will be collected about 5 weeks before any treatment, just before first HER2 BATs infusion, before HER2 BATs #5, before HER2 BATs #8, and 2 weeks, 1 month, 3 months, and 6 months after last Pembrolizumab
  Sequential monitoring of phenotype, IFN-γ EliSpots, anti-breast cancer cytotoxicity of peripheral blood mononuclear cells (PBMC) directed at breast cancer cell lines, Th1/Th2 serum cytokine patterns, and anti-breast cancer antibodies in the serum during the "vaccinate and consolidate" process
Disease control rate | Imaging will be done prior to study treatment, 1 month, 3 months and 6 months after completion of study treatment. Imaging will then be performed according to standard of care.
  The percentage of subjects who achieve complete response, partial response and stable disease following treatment.
Objective response rate | Imaging will be done prior to study treatment, 1 month, 3 months and 6 months after completion of study treatment. Imaging will then be performed according to standard of care.
  The percentage of subjects with a response of complete response (CR) or partial response (PR) per immune related response criteria (irRC)
Duration of response | Imaging will be done prior to study treatment, 1 month, 3 months and 6 months after completion of study treatment. Imaging will then be performed according to standard of care.
  The time from documentation of tumor response to disease progression.
Survival | Every 3 months following last study visit until death or for 10 years
  Progression-free and Overall Survival in a dose-expansion cohort of an additional 12 subjects

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Dillon, MD, Principal Investigator — University of Virginia
Locations (1):
- Ashley Donihee, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lum LG, Thakur A, Al-Kadhimi Z, Colvin GA, Cummings FJ, Legare RD, Dizon DS, Kouttab N, Maizel A, Colaiace W, Liu Q, Rathore R. Targeted T-cell Therapy in Stage IV Breast Cancer: A Phase I Clinical Trial. Clin Cancer Res. 2015 May 15;21(10):2305-14. doi: 10.1158/1078-0432.CCR-14-2280. Epub 2015 Feb 16. PMID 25688159
- [Background] Vaishampayan U, Thakur A, Rathore R, Kouttab N, Lum LG. Phase I Study of Anti-CD3 x Anti-Her2 Bispecific Antibody in Metastatic Castrate Resistant Prostate Cancer Patients. Prostate Cancer. 2015;2015:285193. doi: 10.1155/2015/285193. Epub 2015 Feb 23. PMID 25802762